CLINICAL TRIAL: NCT01920022
Title: Early Versus Delayed Insertion of Nexplanon® at Medical Abortion - a Randomized Controlled Equivalence Trial.
Brief Title: Quickstart of Nexplanon® at Medical Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Gemzell Danielsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QW2013
Record Dates: First submitted 2013-08-06; First posted 2013-08-09 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Early Pregnancy Termination; Medical Abortion; Postabortion Contraception
Keywords: medical abortion; postabortion contraception; LARC; Nexplanon; subdermal contraceptive implant
MeSH Terms: interventions — Mifepristone; etonogestrel; Contraceptive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etonorgestrel and mifepristone (Experimental): Quickstart, insertion of Nexplanon on the day of mifepristone in medical abortion
  Interventions: Drug: Mifepristone; Drug: etonorgestrel
- mifepristone (Active Comparator): Mifepristone on day 1. Nexplanon insertion at 3 weeks FU after the medical abortion
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Day one of medical abortion
Drug: etonorgestrel
  Other Names: Nexplanon, Contraceptive implant
  Arms: Etonorgestrel and mifepristone

SUMMARY:
Women having abortions are at high risk for subsequent unintended pregnancy and repeat abortion. Clearly, encouraging contraceptive use after abortion is a high priority. Long acting reversible contraceptives (LARCs, Implants and intrauterine contraception) are the most effective methods to help women avoid a repeat unwanted pregnancy and abortion. Studies in surgical abortion patients, show that "quickstart" of a LARC - i.e., inserting it during the surgical procedure - is associated with substantially greater use of that method six months later than requiring women to return later to get the device. However, today a majority of women chose medical abortion. The clinical routine is to insert LARCs at the follow up 2 to 3 weeks after the abortion treatment. Frequently women choose to do part of the abortion treatment at home and do not return for a follow up. Thus, the possibility to quick start a contraceptive method in medical abortion would be a major advantage especially if this could be done at the time of administration of mifepristone.

ELIGIBILITY:
Inclusion Criteria:

* women opting for medical abortion and post abortion Nexplanon
* no contraindicated to medical abortion or Nexplanon (according to the SMPc) gestational length up to and including 63 days (determined with ultrasonography)
* able and willing to provide informed consent

Exclusion Criteria:

* unwilling to participate,
* unable to communicate in Swedish and English and
* minors (i.e. women < 18 years of age),
* contraindications to Nexplanon®
* women with pathological pregnancies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 551 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Complete abortions without surgical intervention | at 3 weeks follow up
  Efficacy of the medical abortion treatment

SECONDARY OUTCOMES:
Unplanned pregnancy | during one year FU
  Numbers of pregnancies within the first year following the index abortion
Number of women with complications | evaluated at the 3weeks FU
  reports and rates of AE/SAE
Rate of implant insertion | up to 1year FU
  Compliance, contraceptive usage
Bleeding | Evaluated at 1 year FU
  Bleeding will be evaluated with regard to both bleeding during the medical abortion and bleeding patterns during the one year FU

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Gemzell-Danielsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (7):
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset/Östra, Gothenburg
  - Universitetssjukhuset, Linköping
  - Universitetssjukhuset i Örebro, Örebro
  - Karolinska Universitetssjukhuset, Stockholm
  - Danderyds Hospital, Stockholm
  - Södersjukhuset, Stockholm
- Chalmers Sexual and Reproductive Health Service, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Hognert H, Kopp Kallner H, Cameron S, Nyrelli C, Jawad I, Heller R, Aronsson A, Lindh I, Benson L, Gemzell-Danielsson K. Immediate versus delayed insertion of an etonogestrel releasing implant at medical abortion-a randomized controlled equivalence trial. Hum Reprod. 2016 Nov;31(11):2484-2490. doi: 10.1093/humrep/dew238. Epub 2016 Sep 22. PMID 27664217